CLINICAL TRIAL: NCT01385137
Title: S0927: A Randomized Placebo-Controlled Trial of Omega-3-Fatty Acid for the Control of Aromatase Inhibitor-Induced Musculoskeletal Pain and Stiffness In Women With Early Stage Breast Cancer, Phase III
Brief Title: S0927:Omega3-Fatty Acid Supp in Treating Muscle&Bone Pain&Stiffness in Pts W/Stg I,II,III Brst Canc Rec'v Hormone Thpy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: S0927; S0927 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Arthralgia; Breast Cancer; Pain
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; pain; arthralgia
MeSH Terms: conditions — Arthralgia; Breast Neoplasms; Pain | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral omega-3-fatty acid twice daily (BID) or three times daily (TID) for 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: omega-3 fatty acid
- Arm II (Placebo Comparator): Patients receive oral placebo BID or TID for 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: An omega-3 fatty acid-enriched nutritional supplement may help improve muscle and bone pain and stiffness caused by hormone therapy in patients with breast cancer.

PURPOSE: This randomized phase III trial is studying omega-3 fatty acid supplements in treating muscle and bone pain and stiffness in patients with stage I, stage II, or stage III breast cancer receiving hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether omega-3-fatty acid as compared to placebo causes a reduction in worst joint pain and/or stiffness at 12 weeks, as measured by the modified Brief Pain Inventory (BPI), in women with early-stage breast cancer and aromatase inhibitor (AI)-associated arthralgia.

Secondary

* To assess the proportion of patients who report improved versus deteriorated joint pain with omega-3-fatty acid versus placebo.
* To assess the proportion of patients who report improved versus deteriorated joint stiffness with omega-3-fatty acid versus placebo.
* To assess whether patients receiving omega-3-fatty acid compared to placebo have decreased analgesic use and increased AI adherence.
* To assess whether patients receiving omega-3-fatty acid compared to placebo have improved functioning, pain, and stiffness in the knees/hips (as measured by the Western Ontario and McMaster Universities Osteoarthritis, WOMAC) score.
* To assess whether patients receiving omega-3-fatty acid have improved functioning, pain, and stiffness in the hands (as measured by the Modified Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands, M-SACRAH).
* To assess whether patients receiving omega-3-fatty acid compared to placebo have improved functional quality of life as measured by the Functional Assessment of Cancer Therapy-Endocrine Subscale (FACT-ES) Trial Outcome Index (TOI).
* To assess whether patients receiving omega-3-fatty acid report changes for the better versus worse compared to placebo as measured by the Global Rating of Change Scale.
* To identify minimally important change in the WOMAC, M-SACRAH, and the FACT-ES Trial Outcome Index (TOI) using "a little better" or "a little worse" responses on the patient-reported global rating of change in joint pain and joint stiffness.
* To assess whether patients receiving omega-3-fatty acid compared to placebo have an improved lipid profile as measured by triglycerides, HDL, and LDL.
* To assess the toxicity of omega-3-fatty acid compared to placebo in this setting.
* To assess whether there is a difference in serum-free and total estradiol levels before and after treatment with omega-3-fatty acid compared to placebo.
* To explore whether CYP19A1 genotype correlates with severity of joint symptoms or predicts response to omega-3-fatty acid. (exploratory)
* To explore changes in hormonal and inflammatory serum biomarkers, such as IL6, TNF-α, and CRP.
* To assess whether there is a relationship between change in serum docosahexaenoic acid (DHA) and EPA and resolution of joint symptoms.
* To establish a cohort of patients (placebo group) to better characterize the natural history of the syndrome.

OUTLINE: This is a multicenter study. Patients are stratified according to prior osteoarthritis (yes vs no) and prior taxane use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral omega-3-fatty acid twice daily (BID) or three times daily (TID) for 24 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo BID or TID for 24 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and at 12 and 24 weeks for biomarker and DNA analysis.

Patients complete the Brief Pain Inventory Short Form (BPI-SF), the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index, the Modified-Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH), the FACT-ES Trial Outcome Index, and the Omega-3-fatty acid Dietary Intake questionnaires at baseline and at 6, 12, and 24 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive adenocarcinoma of the breast

  * Stage I, II, or IIIA disease
  * No metastatic disease
* Must have undergone modified radical mastectomy or breast-sparing surgery and recovered
* Estrogen-receptor positive (ER+) and/or progesterone-receptor positive (PR+)
* Currently taking a third-generation aromatase inhibitor (AI) [e.g., anastrozole (Arimidex®), letrozole (Femara®), or exemestane (Aromasin®)] for ≥ 90 days prior to registration with plans to continue for ≥ 180 days after registration
* Must have completed the S092 Brief Pain Inventory (BPI)-Short Form within the past 14 days, and must have a worst pain/stiffness of ≥ 5 on the BPI (item #2) that has started or increased with AI therapy

PATIENT CHARACTERISTICS:

* Postmenopausal
* Zubrod performance status 0-2
* Willing to submit blood for serum-free estradiol, total estradiol, serum inflammatory markers (IL6, TNF-α, CRP), DHA and EPA, lipid profile (LDL, HDL, triglycerides), and DNA analysis (CYP19A1)
* Able to complete study questionnaires in English
* At least 5 years since other malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, ductal carcinoma in situ of the breast or adequately treated stage I or II cancer from which the patient is currently in complete remission
* Patients must not have a known allergy to soy, given that the placebo is suspended in soybean oil

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 months since prior omega-3 fatty acid supplements and must agree to refrain from omega-3-fatty acid supplements from sources outside of this study
* More than 28 days since prior investigational agents
* No other medical therapy, alternative therapy, or physical therapy for joint pain/stiffness within the past 30 days
* Patients must not be on anticoagulation medication (i.e., heparin/warfarin) because of increased risk of bleeding within 28 days prior to registration
* Patients must not have a history of bone fracture or surgery of the afflicted knees and/or hands within 6 months prior to registration
* Patients must not be on narcotics within 14 days of registration
* Patients may have received corticosteroid treatment; however, the following criteria apply:

  * Patients must not have received oral or intramuscular corticosteroids within the 28 days prior to registration
  * Patients must not have received intra-articular steroids to the study, or any other, joint within 28 days prior to registration
* Patients must not have received topical analgesics (e.g., capsaicin preparations) to the study joint or any other analgesics (e.g., opiates, tramadol; with the exception of nonsteroidal antiinflammatory drugs (NSAIDs) and acetaminophen) within 14 days prior to registration

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center; Laurence H. Baker, DO, FACOI, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (292):
- United States (292):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Springdale, Rogers, Arkansas
  - Kaiser Permanente Medical Center - Anaheim/Orange County, Anaheim, California
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente Medical Center - Baldwin Park, Baldwin Park, California
  - Kaiser Permanente Medical Center - Bellflower, Bellflower, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente Medical Center - Fontana, Fontana, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Kaiser Permanente Medical Center - Harbor City, Harbor City, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente - Irvine, Irvine, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Kaiser Foundation Hospital - West Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Mercy Cancer Center at Mercy Medical Center, Merced, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Epic Care - Oakland, Oakland, California
  - Kaiser Permanente Medical Group, Panorama City, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Riverside, Riverside, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Kaiser Permanente Medical Cener - Woodland Hills, Woodland Hills, California
  - Kaiser Permanente - Denver, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute at St. Luke's, Twin Falls, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - CHRISTUS Cabrini Cancer Center, Alexandria, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Singh and Arora Hematology Oncology, PC, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Great Lakes Cancer Institute - Lapeer Campus, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Baylor Medical Center at Irving, Irving, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Rocky Mountain Oncology, Casper, Wyoming

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hershman DL, Unger JM, Crew KD, Awad D, Dakhil SR, Gralow J, Greenlee H, Lew DL, Minasian LM, Till C, Wade JL 3rd, Meyskens FL, Moinpour CM. Randomized Multicenter Placebo-Controlled Trial of Omega-3 Fatty Acids for the Control of Aromatase Inhibitor-Induced Musculoskeletal Pain: SWOG S0927. J Clin Oncol. 2015 Jun 10;33(17):1910-7. doi: 10.1200/JCO.2014.59.5595. Epub 2015 May 4. PMID 25940724

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Omega-3-fatty Acid): Patients receive oral omega-3-fatty acid twice daily (BID) or three times daily (TID) for 24 weeks in the absence of disease progression or unacceptable toxicity
- Arm II (Placebo): Patients receive oral placebo BID or TID for 24 weeks in the absence of disease progression or unacceptable toxicity
Period: Evaluable at Baseline
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Started (9 patients on arm 1 and 4 patients on arm 2 found ineligible after registration) | 131 | 131
Completed | 122 | 127
Not Completed | 9 | 4
Period: Evaluable for Primary Endpoint
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Started | 131 | 131
Completed | 102 | 107
Not Completed | 29 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo) | Total
Number analyzed (Participants) | 122 | 127 | 249
Age, Continuous [Median (Full Range); unit: years] | 59.5 [40 to 84] | 59.1 [43 to 83] | 59.2 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 127 | 249
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 112 | 113 | 225
  Unknown or Not Reported | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 113 | 104 | 217
  Black | 5 | 15 | 20
  Asian | 1 | 3 | 4
  Native American | 0 | 1 | 1
  Multiracial | 1 | 1 | 2
  Unknown | 2 | 3 | 5
Osteoarthritis [Count of Participants; unit: Participants]
  Yes | 28 | 29 | 57
  No | 94 | 98 | 192

OUTCOME MEASURES:

1. Primary Outcome: Week 12 Brief Pain Inventory (BPI) Worst Pain/Stiffness Score
Description: Linear regression model-adjusted week 12 mean score by treatment group.
  Purpose: To assess the severity of pain Population: Patients with pain from chronic diseases or conditions such as cancer, osteoarthritis and low back pain, or with pain from acute conditions such as postoperative pain Responsiveness: Responds to both behavioral and pharmacological pain interventions Method: Self-report or interview Scoring: Higher scores indicate more pain Range: 0-10
Time Frame: 12 weeks post-registration
Measure: Mean (95% Confidence Interval); unit: BPI score
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 102 | 107
BPI score | 5.3 [4.68 to 5.91] | 5.47 [4.86 to 6.09]
Statistical Analysis 1: Comparison: Arm I (Omega-3-fatty Acid) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.58, Regression, Linear; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.79 to 0.44]

2. Secondary Outcome: Number of Patients With Adverse Events That Are Possibly, Probably or Definitely Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 25 weeks
Population: All participants receiving at least some protocol treatment
Measure: Number; unit: Participants
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 117 | 124
Participants
  Arthralgia | 0 | 1
  Diarrhea | 1 | 0
  Dyspepsia | 1 | 0
  Pain | 0 | 1
  Pain in extremity | 1 | 0
  Peripheral motor neuropathy | 0 | 1
  Rash maculo-papular | 0 | 1

3. Secondary Outcome: Week 12 Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score
Description: Linear regression model-adjusted week 12 mean score by treatment group The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores indicate higher symptom burden.
Time Frame: 12 weeks post-registration
Measure: Mean (95% Confidence Interval); unit: WOMAC score
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 102 | 107
WOMAC score | 34.5 [29.4 to 39.7] | 36.7 [31.5 to 41.8]
Statistical Analysis 1: Comparison: Arm I (Omega-3-fatty Acid) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.42, Regression, Linear; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-7.30 to 3.04]

4. Secondary Outcome: Week 12 Modified Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH) Score
Description: Linear regression model-adjusted week 12 mean score by treatment group. Higher scores represent higher symptom burden. Range is 0 to 100.
Time Frame: 12 weeks post-registration
Measure: Mean (95% Confidence Interval); unit: M-SACRAH score
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 100 | 107
M-SACRAH score | 28.8 [23.9 to 33.7] | 28.1 [23.2 to 33]
Statistical Analysis 1: Comparison: Arm I (Omega-3-fatty Acid) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.77, Regression, Linear; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-4.17 to 5.60]

5. Secondary Outcome: Week 12 Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) Score
Description: FACT-ES measures physical, social and family, emotional, and functional well-being and endocrine symptoms. The FACT scaleshave five response levels ("not at all" to "very much"), where higher scores reflect better well-being and fewer symptoms. This scale provided a measure of the broader impact of join pain and stiffness symptoms. Score range is 0 to 220.
Time Frame: 12 weeks post-registration
Measure: Mean (95% Confidence Interval); unit: FACT-ES score
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Number analyzed (Participants) | 100 | 107
FACT-ES score | 95 [91.7 to 98.3] | 92.8 [89.5 to 96.1]
Statistical Analysis 1: Comparison: Arm I (Omega-3-fatty Acid) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.21, Regression, Linear; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [-1.16 to 5.44]

ADVERSE EVENTS:
Time Frame: Up to 25 weeks
Arm/Group | Arm I (Omega-3-fatty Acid) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/124
Other Adverse Events (participants affected / at risk) | 70/117 | 74/124
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Omega-3-fatty Acid) (N=117) | Arm II (Placebo) (N=124)
Bloating (Gastrointestinal disorders) | 7 | 2
Diarrhea (Gastrointestinal disorders) | 18 | 11
Dyspepsia (Gastrointestinal disorders) | 23 | 16
Nausea (Gastrointestinal disorders) | 12 | 17
Fatigue (General disorders) | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 63
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 11 | 15
Headache (Nervous system disorders) | 3 | 7
Hot flashes (Vascular disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No